CLINICAL TRIAL: NCT03612960
Title: Measuring Neuroadaptations in Response to Very Low Nicotine Content Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Andrea Hobkirk, PhD, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 9276; K23DA045081 (NIH)
Record Dates: First submitted 2018-07-18; First posted 2018-08-02 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Dependence
Keywords: Tobacco; Nicotine; Smoking; Functional magnetic resonance imaging; Addiction
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very low nicotine content cigarettes (Experimental): Research cigarettes with very low nicotine content (0.03 mg/cigarette) compared to usual brand cigarettes.
  Interventions: Drug: Very low nicotine content cigarettes
- Normal nicotine content cigarettes (Placebo Comparator): Research cigarettes with normal nicotine content (0.8 mg/cigarette) similar to usual brand cigarettes.
  Interventions: Drug: Normal nicotine content cigarettes

INTERVENTIONS:
Drug: Very low nicotine content cigarettes — Very low nicotine content cigarettes
  Arms: Very low nicotine content cigarettes
Drug: Normal nicotine content cigarettes — Normal nicotine content cigarettes
  Arms: Normal nicotine content cigarettes

SUMMARY:
The overall goal of this study is to determine if switching to very low nicotine content cigarettes changes the function of brain circuitry involved in incentive salience and executive control among dependent smokers.

DETAILED DESCRIPTION:
In a double-blind, randomized controlled trial, dependent smokers will be randomized to a 6-week very low nicotine content (VLNC) cigarette condition (N=50) or a 6-week normal nicotine content cigarette control condition (NNC; N=25). Participants will undergo functional magnetic resonance imaging (fMRI) scans at baseline and 6-weeks to investigate the nicotine-related modulation of brain circuitry involved in incentive salience valuation and executive control. Imaging tasks will engage the incentive salience of smoking cues and non-smoking rewards and executive control functions to identify changes in functional activity within, and effective connectivity between, known salience and executive control brain circuitry. A novel fMRI task using specialized odor presentation equipment and fMRI sequences will assess neural cue reactivity to smoke odors.

ELIGIBILITY:
Inclusion Criteria:

* 21-60 years old
* Smoke >5 cigarettes per day
* >1 year of daily smoking
* No quit attempt in prior month and not planning to quit smoking within next 3 months
* Able to understand and consent to study procedures
* High school or lower educational attainment or annual household income < $50,000
* Plan to live in local area next 3 months
* Women not pregnant or nursing and taking steps to avoid pregnancy
* Able to read and write in English
* Access to computer with internet service that allows for Zoom

Exclusion Criteria:

* Use of non-cigarette tobacco products in the past 7 days
* Use of illicit substances more than once a week in the past 3 months (excluding marijuana)
* Current alcohol abuse impairing participation
* MRI safety contraindications (e.g., metal implants, claustrophobia)
* Unstable or significant medical conditions (e.g., chronic obstructive pulmonary disorder, coronary heart disease)
* Major neurological conditions or brain trauma
* Major surgeries planned in next 3 months
* Use of smoking cessation medication in prior month (e.g., varenicline, patch)
* Uncontrolled serious mental illness, suicidality, or inpatient psychiatric hospitalization in the past 6 months
* Unwillingness to provide urine samples
* Unwilling to smoke study assigned cigarettes for the remainder of the trial
* Plans to move or take extended travel out of the area in the next 3 months
* Any other condition or situation that would, in the investigator's opinion, make it unlikely that the participant could comply with the study protocol
* Self-reported color blindness
* Left-handedness
* Smell dysfunction as determined via standardized assessment

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hobkirk, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Started | 21 | 13
Completed | 20 | 10
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 21 | 13 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.90 (7.98) | 44.46 (8.69) | 43.50 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 13 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 12 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 13 | 34
Cigarettes per day (CPD) [Mean (Standard Deviation); unit: cigarettes per day] — Cigarettes per Day at Baseline
  cigarettes per day | 18.90 (7.35) | 14.46 (5.39) | 17.21 (7.01)
Menthol vs Non-Menthol [Count of Participants; unit: Participants] — Menthol vs Non-Menthol Cigarettes smoked at baseline
  Participants
    Menthol | 15 | 6 | 21
    Non-Menthol | 6 | 7 | 13
Cigarette Dependence [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom Test for Cigarette Dependence score at baseline. Scores range from 0 to 10, with 10 indicating higher dependence on cigarettes.
  units on a scale | 4.10 (1.22) | 3.77 (1.09) | 3.97 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Oxygen Level Dependent (BOLD) Signal Collected by Functional Magnetic Resonance Imaging (fMRI) During Monetary Delay Discounting Task
Description: Change from baseline to 6-weeks post-intervention in percentage of BOLD signal during hard vs. no choice conditions on a monetary delay discounting task in a left-sided cortical brain region encompassing the central opercular and dorsolateral prefrontal cortices.
Time Frame: Change in BOLD signal from baseline to the 6-week visit.
Population: Only participants who completed the baseline and post-randomization laboratory visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 20 | 10
Percent change | 0.13 (0.18) | -0.16 (0.18)
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.14 to 0.43], Standard Error of Mean 0.07; The mean percent change in BOLD signal used for this t-test was extracted from a brain cluster with significant group differences in changes in activation over time (voxel p<.05, cluster p<.05) identified using a whole-brain, voxel-wise two-way mixed effect ANOVA with FSL software

2. Secondary Outcome: Change in Self-reported Cigarettes Per Day
Description: Difference in week 6 mean minus week 1 mean of cigarettes used per day reported by participants on daily logs.
Time Frame: Average cigarettes per day during week 1 subtracted from average cigarettes per day during week 6.
Measure: Mean (Standard Deviation); unit: Number of cigarettes per day
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 20 | 10
Number of cigarettes per day | -5.1 (7.9) | 3.3 (16.0)
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p = .063, t-test, 2 sided; Mean Difference (Final Values) = -8.38, 95% CI 2-sided [-17.24 to 0.48], Standard Error of Mean 4.33

3. Secondary Outcome: Change in Percentage of Immediate Choices on Monetary Delay Discounting Task
Description: A difference score (6-weeks minus baseline) of the percentage of trials where the immediate (vs. delayed) monetary option was chosen out of all task trials during the monetary delay discounting task that was completed outside of the MRI scan.
Time Frame: Changes from baseline to 6-weeks post intervention.
Population: Participants who completed both trial laboratory visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in percentage
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 20 | 10
Change in percentage | 0.20 (30.26) | 1.57 (9.16)
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p = 0.890, t-test, 2 sided; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-21.57 to 18.82], Standard Error of Mean 9.86

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/13
Other Adverse Events (participants affected / at risk) | 1/21 | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Nicotine Content Cigarettes (N=21) | Normal Nicotine Content Cigarettes (N=13)
Fractured Finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject fractured their finger at their work, went to urgent care and was treated there. Was determined to not be related to the study.
Nausea and Headaches (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject had more frequent headaches and nausea after starting a new medication around the same time they began using study products.

LIMITATIONS AND CAVEATS:
Exclusion criteria was revised throughout the project (e.g., removed menthol use as exclusion) to accommodate challenges in recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03612960/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03612960/ICF_001.pdf